CLINICAL TRIAL: NCT01263340
Title: Observational, Multi-centre, Retrospective Cohort Study to Evaluate Prevalence, Incidence, Severity, Co-morbidities and Burden of Disease in Patients With a Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) by Close Scrutiny of the Patient Journey
Brief Title: Characterisation of People With COPD
Acronym: CoCO
Status: Completed | Type: Observational
Sponsor: National Services for Health Improvement Ltd (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SCO115217
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; observational study; prevalence; characterisation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- People with COPD

SUMMARY:
The investigators will describe the characteristics, prevalence, incidence, severity co-morbidity and management of patients with chronic obstructive pulmonary disease (COPD) in the UK. 100 practices will be sampled amounting to a total study population of about 10 000 patients. Information will be collected electronically and, where necessary, by a hand search of patient records.

DETAILED DESCRIPTION:
Research questions:

1. What is the recorded prevalence of COPD in the UK? [numerator: the prevalence of COPD defined as ANY current READ code for COPD or inclusion in a COPD register denominator: the whole population]

   * What proportion of this population has documented spirometry to confirm the diagnosis?
   * What proportion has documented spirometry in the last year?
   * What proportion has ever had a documented history of asthma?
   * What proportion currently has a documented history of asthma?
   * What proportion currently smokes?
   * What proportion of smokers has a record of receiving smoking cessation advice?
   * What proportion of smokers has had a prescription for smoking cessation therapy?
   * What proportion of people with COPD has a READ code for exception reporting?
   * What are their demographic features? (height weight, BMI, age, smoking status, forced expiratory flow in 1st second (FEV1_, DOSE)
   * What proportion of people with COPD has a READ code for exception reporting from spirometry?
   * What are their demographic features? (height, weight, body mass index (BMI), age, smoking status, FEV1, DOSE)

   Sub analysis: descriptions and comparison of prevalence by • Age

   • geographical location of participating practices

   • primary care training practice

   • number of performing general practitioners (GPs) in practice (<3 v >/= 3)
2. What is the incidence of COPD in the UK

   • number of people with a new diagnosis of COPD in the last year as a proportion of the whole population
3. What is the distribution of severities of COPD?

   • Description of severity of airflow obstruction by FEV1 measurement:

   Mild (FEV1 ≥ 80% predicted):

   Moderate (FEV1 50% to 79% predicted) Severe (FEV1 30% to 49% predicted) Very severe (FEV1 ≤ 30% predicted)

   • And by DOSE

   Compare the severity of disease (exacerbation rate) according to DOSE "high risk" and "low risk" and compare this to the stratification of severity in the study population by degree of airflow limitation.

   • And by COPD Assessment Test (CAT)

   Explore the use of CAT in clinical practice and the availability and spread of data
4. What is the exacerbation rate?

   * In the last year in people with a diagnosis of COPD > 1 year
   * In the last three years in people with a diagnosis of COPD > 3years (as a proportion of the population with COPD).
   * What is the seasonal variation of COPD exacerbations: what proportion of exacerbations occurs in each month of the year?
   * Do recurrent primary care managed exacerbations predict hospital admissions? What is the prior exacerbation rate in patients admitted to hospital? Population of interest: those with hospital admissions for COPD: what is the exacerbation rate (and time frame of exacerbations) prior to a hospital admission?

     4a. What proportion of the COPD population had at least one exacerbation?

   Hospital attendance: Any documented visit to any secondary care (not primary care out of hours) site with no overnight stay

   Hospital admission: Any documented visit to any secondary care site with an overnight stay with a principal diagnosis of COPD or chest infection or pneumonia or exacerbation of asthma ICU admission: Any documented admission to any high dependency unit (note, AN EXPLORATORY EXERCISE. Validity of this data in primary care record is questionable)

   Death: Any death with COPD documented as the primary cause or within 14 days of the onset of an exacerbation (EXPLORATORY)
   * Does DOSE predict undesirable outcomes (death, hospital admission, exacerbation rate)?
   * Does FEV1 predict undesirable outcomes (death, hospital admission, exacerbation rate)?
   * Does medical research council dyspnoea (MRC) score (or other component of DOSE) predict undesirable outcomes?
   * Possible exploratory analysis: does ADO index (Age, Dyspnoea (MRC score) Obstruction (FEV1 % pred)) predict undesirable outcomes?
   * Does number of patients in a practice receiving a Tiotropium prescription predict hospital admission at a practice level?
5. Therapy:

   * What proportion of patients (without a diagnosis of asthma) receives inhaled glucocorticosteroids at unlicensed doses (any steroid (fluticasone, budesonide, beclometasone, ciclesonide) or combination Seretide, Symbicort, Fostair) EXCEPT Seretide Accuhaler 50/500 or Symbicort?
   * What proportion of patients with FEV1> 50 and no diagnosis of asthma receive any steroid preparation? (Note: Seretide Accuhaler 50/500 is licensed for use in patients with COPD and (pre-bronchodilator) FEV1 < 60% predicted and is therefore not subject to off label use in this instance). The approach outlined here is a consensus for the purposes of identifying a pragmatic approach to data collection.
   * What proportion of patients with FEV<50 do not receive any inhaled steroid?
   * What proportion of patients with 1 or more exacerbation in the last year does not receive any inhaled steroid?
   * What proportion of patients with FEV1 <50 do not receive Seretide 50/500 or Symbicort?
   * What proportion of patients are on "triple therapy" i.e. Seretide or Symbicort PLUS Tiotropium, classified by severity (FEV1)
   * What is the refill rate for prescriptions by class (all above and SABA) in the previous year?
   * What proportion of patients have an MRC dyspnoea score >/= 3?
   * What proportion of these patients has been referred for pulmonary rehabilitation?
   * What proportion has received pulmonary rehabilitation?
   * What proportion has documented evidence of receiving a self management plan?
6. Co-morbidities:

   What proportion of patients with COPD have any READ code ever for the following co-morbidities:
   * Cardiovascular disease
   * Cerebrovascular disease
   * Diabetes Mellitus
   * Cancer
   * Lung cancer
   * Depression
   * Osteoporosis What proportion of patients with at least one comorbidity has attended a specialist chest service / clinic in the last year? What is the exacerbation rate in this group v patients without comorbidity? What is the hospital admission rate in this group v the rest? What proportion of the population has a record of NEVER smoking? What are the features of this group (age, sex, geography, exacerbation rate, medication, comorbidities
7. Newly diagnosed patients

   * What are the characteristics (demographics: height weight, BMI, age, smoking status, FEV1, DOSE) of newly diagnosed patients (first READ code for COPD within the last year)?
   * What proportion of these patients received a prescription for Tiotropium within 1 month of diagnosis?
   * What proportion of these patients received a prescription for an inhaled corticosteroid / longa acting beta-agonist fixed dose (ICS / LABA) combination within 1 month of diagnosis?
   * In patients FEV1 <50% predicted, what proportion receive a) Tiotropium and b) an ICS / LABA combination first
   * What proportion of these patients with FEV1>50 received a prescription for ICS / LABA combination within 1 month of diagnosis?
8. General Practice Research database (GPRD)

   * What proportion of our sample currently contributes to the GPRD database?
   * Are their differences in the features of the two groups: Age geographical location of participating practices, primary care training practice, number of performing GPs in practice (<3 v >/= 3), disease severity (DOSE, FEV1) exacerbation rate
9. What changes have there been at practice level to the above parameters in the last year?

ELIGIBILITY:
Inclusion Criteria:

* people with a read code diagnosis of COPD

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with a Read code diagnosis of COPD
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Prevalence and characterisation of people with COPD | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Haughney, FRCPE FRCGP, Principal Investigator — NSHI Ltd
Locations (1):
- NHS primary care centres, Nationwide, United Kingdom

REFERENCES:
- [Derived] Haughney J, Gruffydd-Jones K, Roberts J, Lee AJ, Hardwell A, McGarvey L. The distribution of COPD in UK general practice using the new GOLD classification. Eur Respir J. 2014 Apr;43(4):993-1002. doi: 10.1183/09031936.00065013. Epub 2013 Oct 31. PMID 24176990